CLINICAL TRIAL: NCT05368922
Title: Upper Limb Rehabilitation Using Virtual Reality in Children With Cerebral Palsy
Brief Title: Upper Limb Rehabilitation Using Virtual Reality in Children With Cerebral Palsy (RV-REEDUC)
Acronym: RV-REEDUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slb Pharma (Other)
Collaborators: European Regional Development Fund (Other); La Région Basse-Normandie (Other); Université de Caen Normandie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV-Reeduc
Record Dates: First submitted 2022-04-19; First posted 2022-05-10 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy; Brain Diseases
Keywords: Cerebral Palsy; Virtual Reality; Immersive Virtual Reality; Rehabilitation; Upper Limb; Upper extremity
MeSH Terms: conditions — Cerebral Palsy; Brain Diseases

STUDY DESIGN:
Intervention Model Description: A multi-center randomized controlled trial will be implemented across three different locations. Twenty-two children will be randomly divided into an experimental group that will follow a virtual reality rehabilitation protocol with a pre-test and two post tests and with three weekly sessions for four weeks, and a control group which will only carry out the pre and posttests.
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Virtual Reality Group (Experimental): Children will receive a virtual reality rehabilitation protocol for their most affected upper limb for four weeks, on the basis of three sessions a week, in addition to their usual care. Virtual reality will be applied to participants for 30 minutes and will be based on two perceptual-motor tasks.
  Interventions: Device: Virtual reality rehabilitation
- Control group (No Intervention): Children who will be randomized to the control group will follow their usual care for four weeks (usual motor activity, including classical rehabilitation and sports or physical activities). The rehabilitation protocol will be proposed after the second post-test

INTERVENTIONS:
Device: Virtual reality rehabilitation — The virtual reality rehabilitation protocol will be based on two perceptual-motor tasks (e.g., visuomotor tracking task and pointing task) in a 3D environment. The visuomotor tracking task will consist in tracking a virtual target moving with an effector manipulated by a remote controller. The pointing task will consist in tapping targets that are in a cube as quickly as possible with an effector manipulated by a remote controller. Both tasks will be performed in a 3D virtual playful environment.
  The rehabilitation protocol will follow a progression through the manipulation of the virtual environment and the constraints of the tasks.
  Arms: Experimental: Virtual Reality Group

SUMMARY:
This study aims to evaluate the effect of a virtual reality rehabilitation protocol on visuo-motor coordination and upper limb functional abilities in children with unilateral or bilateral cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is the most common cause of motor disability in childhood. Motor disorders result in significant upper limb impairments involving limitations in daily activities. Functional rehabilitation of the upper limb therefore appears to be of primary importance in the management of this condition. However, conventional rehabilitation programs encounter some limitations such as the repetitiveness and the lack of attractivity of the proposed protocols and the poor transfer in activities of daily life. In this context, virtual reality appears as a promising tool to provide more attractive and playful protocols with a better control and a better progressivity in the stages of rehabilitation. However, scientific evidence in this area is still insufficient to define and validate specific and safe rehabilitation programs. The goal of this study is to evaluate the effects of a virtual reality rehabilitation protocol on the improvement of visuo-motor coordination and functional abilities in children with cerebral palsy. This study will include twenty-two children with unilateral or bilateral cerebral palsy who will be randomly divided into two groups: one group receiving three weekly virtual reality rehabilitation sessions for four weeks, in addition to their usual activities, and a control group only following its usual care in the same period (classical rehabilitation). Participants will be randomly matched for age, type of cerebral palsy, (hemiplegia, quadriplegia or monoplegia) and the Manual Ability Classification System (MACS). The effectiveness of the rehabilitation protocol will be evaluated through several tests assessing motor functions of the upper limb. Thus, the visuo-motor coordination, manual dexterity, evolution of joint amplitudes, kinematics of movements and functional use of the affected upper limb in daily tasks will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 16 years old,
* Diagnosed as spastic, dyskinetic or ataxic cerebral palsy,
* Diagnosed as hemiplegia, quadriplegia or monoplegia of the upper limb,
* Child without an intellectual disability or with a mild or moderate disability
* Ability to understand the task by to follow verbal instructions,
* Child who has agreed to participate in the study,
* Child whose parents and/or legal guardians have given their consent for his/her participation in the study
* Child who can voluntarily move his affected upper limb in a sufficient range of motion
* Child who is a beneficiary of social security system

Exclusion Criteria:

* Child with epilepsy
* Diagnosed as diplegia or monoplegia of lower limb,
* Severe or profound intellectual disability,
* Severe attention deficit,
* Pain on mobilizing upper limb
* Botulinum toxin injections or surgery on the upper limb within 4 months of the experiment,
* Health condition not allowing participation in the study protocol,
* Pregnant participant,
* Simultaneous participation in another clinical research

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change in visuomotor coordination measured by the "Drawing Trail item" of the manual dexterity domain on Movement Assessment Battery for Children | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  The test measures the number of failures (number of times the boundaries are crossed) performed when tracing a continuous line on a trail. A decrease in the number of failures means a better performance
Change in speed and accuracy of movement measured by the " Posting coins item" of the manual dexterity domain on Movement Assessment Battery for Children | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  The test measures the time needed in seconds to posting 6 coins into a money box with the affected hand. A lower time means a better performance
Change in bimanual coordination measured by the "Threading beads item" of the manual dexterity domain on Movement Assessment Battery for Children | Time frame: Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  The test measures the time needed in seconds to threading 6 beads onto a string. A lower time means a better performance

SECONDARY OUTCOMES:
Change in performance measured by the "Catching Beanbag item" of the Aiming and Catching domain on Movement Assessment Battery for Children | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  The test measures the quantity of bags caught with both hands, thrown by the tester from a distance of 1.80m. Score ranges from 0-10 correct attempts (bags). A higher number of bags caught means a better performance
Change in performance on the " Throwing Beanbag on to Mat item" of the Aiming and Catching domain of Movement Assessment Battery for Children | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  The test measures the quantity of bags throw on to mat. Score ranges from 0-10 correct attempts (bags). A higher number of bags hit means better performance.
Change in manual dexterity measured by the Box and Block Test | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  The test measures the number of transported blocks from one compartment of a box to another of equal size, within 60 seconds. Score ranges from 0-150 blocks. A higher number of blocks means better performance
Change on score of Children's Hand-use Experience Questionnaire (27 questions) | Pre-test (week 1), post-test (at 6 weeks) and 3 months follow-up (at 18 weeks)
  The questionnaire evaluates the experience of children in using the hand, with decreased function, in activities where usually two hands are needed. Score ranges from 0-100). A higher score means a better use of the hand in daily activities
Change in Range of Motion Measurement of upper extremity | Pre-test (week 1), post-test (at 6 weeks) and 3 months follow-up (at 18 weeks)
  Goniometric measurements of upper extremity range of motion (shoulder and elbow) will be done actively
Change in distance-to-target score measured by a visuomotor tracking task performed in virtual reality | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  The score is measured in meters (m). A lower score means a better performance
Change in target contact time score measured by a visuomotor tracking task performed in virtual reality | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  Score ranges from 0-100 and is measured in percent. A higher score means a better performance
Change in elbow joint range of motion measured by a visuomotor tracking task performed in virtual reality | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  Range of motion is measured in degrees. An increase in range of motion means a better outcome
Change in fluidity of movement score measured by a visuomotor tracking task performed in virtual reality | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  Fluidity of movement is measured in with the jerk in m/s3. A lower score means a better outcome
Change in movement time score measured by a pointing task performed in virtual reality | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  The movement time is measured in seconds. A lower score means a better outcome
Change in reaction time score measured by a pointing task performed in virtual reality | Pre-test (week 1), post-test (at 6 weeks), 3 months follow-up (at 18 weeks)
  The reaction time is measured in seconds. A lower score means a better outcome
Intrinsic Motivation Inventory (IMI) | Pre-test ( week 1), post-test (at 6 weeks) and at the sixth session of virtual reality rehabilitation protocol
  Change on score of IMI - adapted version (12 questions)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Benguigui, Pr, Principal Investigator — University of Caen Normandy
Locations (3):
- France (3):
  - Institute of Motor Education (IEM) François Xavier Falala, Hérouville-Saint-Clair, Normandy
  - Physical Medicine and Rehabilitation Center for Children and Adolescent La Clairière, Hérouville-Saint-Clair, Normandy
  - E.P.A Helen Keller, Le Havre, Normandy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burin-Chu S, Baillet H, Leconte P, Lejeune L, Thouvarecq R, Benguigui N. Effectiveness of virtual reality interventions of the upper limb in children and young adults with cerebral palsy: A systematic review with meta-analysis. Clin Rehabil. 2024 Jan;38(1):15-33. doi: 10.1177/02692155231187858. Epub 2023 Jul 27. PMID 37499213